CLINICAL TRIAL: NCT01942239
Title: Real-time Continuous Glucose Monitoring Reduces Duration of Hypoglycemia Episodes in Very Low Birth Weight Neonates
Brief Title: Real-time Continuous Glucose Monitoring in Very Low Birth Weight Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RT-CGMS
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hypoglycemia
Keywords: hypoglycemia; very low birth weight neonate; continuous glucose monitoring
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGM-group (Active Comparator): CGM-group: the intervention(s) to be administered is Continuous glucose monitoring with real time glycemia each 5 minutes
  Interventions: Device: real time continuous glucose monitoring
- IGM-group (No Intervention): IGM-group: the intervention(s) to be administered is intermittent capillary glucose testing (IGM-group) associated with a blind-CGMS to detect retrospectively missed hypoglycemia

INTERVENTIONS:
Device: real time continuous glucose monitoring
  Arms: CGM-group

SUMMARY:
Hypoglycemia is frequent in very low birth weight (VLBW) neonates and compromises their neurological outcome. The aim of this study was to compare real-time continuous glucose monitoring system (RT-CGMS) to standard method by intermittent capillary blood glucose testing in detecting and managing hypoglycemia. The investigators calculated a number of 48 neonates to be randomized between 2 ways of glucose level monitoring for their 3 first days of life : either by RT-CGMS (CGM-group), or by intermittent capillary glucose testing (IGM-group) associated with a blind-CGMS to detect retrospectively missed hypoglycemia. The investigators' hypothesis is that in the CGM group number and duration of hypoglycemia will be lower.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight (VLBW) preterm infants (birth weight under 1500g) who were admitted before 24 hours of life in the Department of Neonatology of the University Hospital of Tours

Exclusion Criteria:

* a serious congenital abnormality,
* a skin condition that contraindicated continuous glucose monitoring,
* a transfer toward another hospital during the first days of life
* an absence of parental agreement.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
number of hypoglycemia episodes | at the end of the first 3 days of life
  hypoglycemia was defined as interstitial glucose level <50 mg/dl; consecutive or <30 min data points <50 mg/dl were defined as a single episode of low glucose concentration.

SECONDARY OUTCOMES:
duration of hypoglycemic episodes | after their 3 first days of life
  hypoglycemia was defined as interstitial glucose level <50 mg/dl. Consecutive or <30 min data points <50 mg/dl were defined as a single episode of low glucose concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Aude Chemin, MD, Principal Investigator — UH Tours
Locations (1):
- UH Tours Clocheville hospital, Tours, France

REFERENCES:
- [Result] Uettwiller F, Chemin A, Bonnemaison E, Favrais G, Saliba E, Labarthe F. Real-time continuous glucose monitoring reduces the duration of hypoglycemia episodes: a randomized trial in very low birth weight neonates. PLoS One. 2015 Jan 15;10(1):e0116255. doi: 10.1371/journal.pone.0116255. eCollection 2015. PMID 25590334